CLINICAL TRIAL: NCT01846364
Title: Diindolymethane: Anti-proliferation Agent in Thyroid Disease-Non-surgical Protocol
Brief Title: DIM as a Treatment for Thyroid Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of sufficient enrollment
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Stimpson P. Schantz, Principal Investigator, The New York Eye & Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NYEEI06.33
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Proliferative Thyroid Disease
Keywords: Thyroid; DIM
MeSH Terms: conditions — Thyroid Diseases | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Subjects with proliferative thyroid disease
  Interventions: Dietary Supplement: Diindolylmethane (DIM)

INTERVENTIONS:
Dietary Supplement: Diindolylmethane (DIM) — 300 mg of Bioresponse DIM (100mg/day of active DIM) a day for 30 days

SUMMARY:
Diindolylmethane (DIM), a dietary supplement, found naturally in cruciferous vegetables (such as cabbage, cauliflower, broccoli, & Brussels sprouts) has been studied extensively in recent years for its anti-cancer effects. DIM has been shown to exert control over cancer cell growth in breast, uterine, cervical, ovarian, and colon cancer.

To date no human study has been published regarding the bioavailability of DIM in thyroid tissue or its effects in proliferative thyroid disease. Our previous study attempted to elucidate DIM's promotion of anti-proliferative estrogen metabolites in proliferative thyroid disease and ascertain its uptake in thyroid tissue. DIM has been shown to concentrate in the thyroid gland. Furthermore, thyroid volumes have been seen to decrease subjectively.

This study would continue our attempt to elucidate DIM's promotion of anti-proliferative estrogen metabolites in proliferative thyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with abnormalities of the thyroid gland suspicious for benign adenoma, or goiterous changes.

Exclusion Criteria:

* Patients who are pregnant, attempting to conceive, or lactating will be excluded due to possible deleterious effects of treatment on fetus/infant. Patients taking oral contraceptives, estrogen therapy, tamoxifin or those with a history of breast cancer will be excluded. Patients with liver disease and those taking statins for hypercholesterolemia will also be excluded to decrease the potential for possible liver toxicity. Any patient with elevated liver enzymes on pretreatment blood screening will be excluded from study participation. Patients with serious systemic diseases such as renal failure, diabetes, blood dyscrasia, coagulopathy, and non-optimized cardiopulmonary disease will be excluded due to the possibility of confounding blood tests screening for toxicity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evidence of objective and quantifiable changes in thyroid size as a resalt of the oral administration of DIM, confirmed by pre- and post- DIM treatment ultrasounds | after 30 days of DIM consumption and 2 and 4 weeks after DIM consumption stopped

SECONDARY OUTCOMES:
Evidence of DIM's effect on estrogen metabolites, confirmed by plasma and urine analysis | after 30 days of DIM consumption

CONTACTS AND LOCATIONS:
Overall Officials: Stimson P. Schantz, MD, Principal Investigator — The New York Eye & Ear Infirmary
Locations (1):
- The New York Eye & Ear Infirmary, New York, New York, United States